CLINICAL TRIAL: NCT06883318
Title: Physical, Psychological and Socioeconomic Effects of Childhood Onset Diabetes in Sweden - Longitudinal Register Based Studies
Brief Title: Physical, Psychological and Socioeconomic Effects of Childhood Onset Diabetes in Sweden
Status: Active, not recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Uppsala University (Other); Lund University (Other); The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-02492
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes Mellitus (T1DM); End-Stage Renal Disease
Keywords: Type 1 diabetes; Childhood-onset; Risk factors; Complications; Socioeconomic conditions
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with childhood-onset type 1 diabetes
- Healthy controls

SUMMARY:
The researchers study time trends of childhood-onset type 1 diabetes and its most serious complication, end-stage renal disease. They further analyse physical, psychological and socio-economic long-term effects on patients and families to identify potentially preventive factors in a population perspective. The researchers investigate the economic burden of disease and study and improve statistical methods for case-control data. The projects use a longitudinal nationwide database involving about 23 000 childhood-onset diabetes cases with maximum follow-up of 48 years and for each case 4 matched controls. The Swedish Childhood Diabetes Register is linked to a number of official, Swedish registers: the Renal register, the Cause of Death register, the National Patient register, the Prescribed Drugs register, the Cancer register and the Integrated Database for Labour Market Research. The researchers use GAM modelling for time trend analyses, standard case-control/cohort analyses, Cox regression for life table analyses, linear fixed effect probability for career development and propensity score models for confounding. The project group is multidisciplinary and involves experts in paediatrics, nephrology, epidemiology, health economics and statistics. This unique database and team continues to yield population-based new knowledge on the consequences of this increasingly common chronic childhood-onset disease.

ELIGIBILITY:
Inclusion Criteria:

* Two prescriptions of insulin in the Prescribed Drug register.
* Age below 15 years of age. Controls are of the same age and born in the same municipality as the cases.

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Swedish Childhood Diabetes Register (SCDR) is based on collaboration with all paediatric clinics in Sweden; from 1977 until 2010 the clinics helped with data collection. Since 2011 the National Board of Health provides new incident data from insulin pre-scriptions using the Prescribed Drug register (PDR). It recruits all cases of type 1 diabetes in children below 15 years. To each case four controls have been assigned through Statistics Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 115000 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of type 1 | From the inception of the data base in July 1977 through 2029
  Incidence of type 1 diabetes in individuals below 15 years of age in Sweden

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Sciences, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No
Data come from official Swedish registers through Statistics Sweden and National Board of Health and Welfare where researchers have access to pseudonymonised information. The ethical permit does not allow sharing of data.

DOCUMENTS (1):
  • Study Protocol (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT06883318/Prot_001.pdf